CLINICAL TRIAL: NCT06969040
Title: Evaluation of the Efficacy of Standard Cognitive Behavioural Therapy + Transcranial Alternating Current in the Treatment of Refractory Insomnia Disorder
Brief Title: The Effect of Standard Cognitive-behavioral Therapy+Transcranial Alternating Current on Refractory Insomnia Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBTI+tACS for TRI
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Insomnia
Keywords: Standard Cognitive Behavioural Therapy; tACS; Treatment-Resistant Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBTI+tACS (Experimental)
  Interventions: Other: CBTI + tACS
- CBTI + Sham tACS (Sham Comparator)
  Interventions: Other: CBTI + Sham tACS

INTERVENTIONS:
Other: CBTI + tACS — CBTI + tACS group method: CBTI for about 50 minutes each time, for a total of 6 weeks: ① first interview: enrolment assessment; ② second interview: treatment initiation; ③ third interview: sleep titration and sleep hygiene; ④ fourth interview: sleep titration; ⑤ fifth-seventh interview: sleep titration; ⑥ eighth interview: sleep titration (end of standardised CBTI treatment. tACS true stimulation) : Transcranial alternating current therapy (tACS) was operated during the same period of CBTI, with 3 electrodes, placed in the prefrontal lobe and bilateral mastoid; the stimulation intensity was 77.5 Hz, 15 mA, 40 min each time, once a day, 5 days a week, for 6 weeks.
  Arms: CBTI+tACS
Other: CBTI + Sham tACS — CBTI+sham tACS group method: CBTI treatment method was the same as before. tACS pseudo-stimulation: the electrode placement position, stimulation frequency, and time settings were the same as the real stimulation, and the stimulation process only had the output of gradual rising and falling current at the beginning and the last 10s, respectively, so as to make the subjects produce the same subjective feelings as the real stimulation.
  Arms: CBTI + Sham tACS

SUMMARY:
The main purpose of this study is to investigate the efficacy of CBTI + transcranial alternating current (TAC) technology in the treatment of refractory insomnia and the mechanism of 'cognitive-behavioural-brain network' interactions.

DETAILED DESCRIPTION:
Difficult to treat insomnia is a sleep disorder that significantly reduces the quality of sleep for patients, seriously affecting their daily work and study. At present, the main treatment method for refractory insomnia in clinical practice is drug therapy. The problems with drug therapy mainly include easy recurrence after discontinuation and the need for long-term or even lifelong medication. However, tolerance or other adverse reactions limit its long-term use. In recent years, studies have shown that cognitive-behavioral therapy and transcranial alternating current stimulation are effective in treating chronic insomnia, prolonging sleep time and improving sleep quality. However, there have been no reports on the efficacy and safety of CBTI combined with tACS in the treatment of refractory insomnia. Based on the important role of tACS in regulating cortical excitability and spontaneous EEG activity, as well as the precise efficacy of CBTI in improving insomnia, we plan to use CBTI combined with tACS to treat refractory insomnia disorders, in order to improve the effectiveness of treatment. This study adopts a randomized double-blind controlled trial to investigate the efficacy and safety of CBT+tACS in the treatment of refractory insomnia, aiming to provide a basis for clinical data of CBT+tACS in the treatment of refractory insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for insomnia in DSM-5;
2. Pittsburgh Sleep Quality Index (PSQI) total score>5 points;
3. Age ≥ 18 years old, with a junior high school education or above;
4. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Individuals with severe physical or mental illnesses are at risk of suicide;
2. Clinically diagnosed or suspected sleep breathing disorders, restless leg syndrome, and sleep wake rhythm disorders, as well as workers on rotating shifts;
3. Pregnant and lactating women;
4. Currently undergoing any psychological therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Differences in change from baseline in Pittsburgh sleep quality index (PSQI) scores at the end of treatment in the two groups | Baseline to week 6

SECONDARY OUTCOMES:
Differences in changes in PSQI scores compared to baseline during follow-up at 3, 6, and 12 months between the two groups | Baseline to week 6, month 3, month 6, and month 12
Differences in the changes in Beck Depression Inventory (BDI) scores from baseline at the end of treatment and follow-up at 3, 6, and 12 months between the two groups | Baseline to week 6, month 3, month 6, and month 12
Differences in Beck Anxiety Inventory (BAI) scores between the two groups at the end of treatment, 3 months, 6 months, and 12 months of follow-up compared to baseline. | Baseline to week 6, month 3, month 6, and month 12
Differences in changes in sleep hygiene awareness and practice scale (SHAPS) between the two groups compared to baseline at the end of treatment, 3 months, 6 months, and 12 months of follow-up [2]. | Baseline to week 6, month 3, month 6, and month 12
Differences in changes in the Insomnia Severity Index (ISI) scores between the two groups at the end of treatment, 3 months, 6 months, and 12 months of follow-up compared to baseline. | Baseline to week 6, month 3, month 6, and month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No